CLINICAL TRIAL: NCT01634906
Title: Erythrocyte-bound Apolipoprotein B After Withdrawal of Statin Therapy
Acronym: EBABAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, Boudewijn Klop, MD, Sint Franciscus Gasthuis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL37698.101.11
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Hyperlipidemia; Atherosclerosis
Keywords: Apolipoprotein B, erythrocytes, statins
MeSH Terms: conditions — Hyperlipidemias; Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Discontinuation of statin therapy (Experimental)
  Interventions: Drug: Temporary discontinuation of statin therapy

INTERVENTIONS:
Drug: Temporary discontinuation of statin therapy — All statins, e.g. atorvastatin, simvastatin, fluvastatin, rosuvastatin, pravastatin
  Other Names: e.g. Crestor, Lipitor

SUMMARY:
Background: preliminary data have shown that erythrocyte-bound apolipoprotein B (ery-apoB) may be protective against atherosclerosis. However, statins may have an effect on ery-apoB.

Objective: to investigate the effect of statins on ery-apoB levels.

Study design: a non-randomized intervention study. Ery-apoB will be measured twice in volunteers who are on statin therapy for medical reasons. After a baseline measurement of ery-apoB volunteers will discontinue their statin use for a period of six weeks followed by a second measurement of ery-apoB. Consecutively subjects will start with their original statin therapy again.

Study population: patients on statin therapy aged 18 years or older.

Intervention: temporary discontinuation of statin therapy for a period of six weeks.

Main study endpoints: changes in ery-apoB levels.

Risks, burden and benefits on participation: volunteers will visit the outpatient clinic twice, the second visit will be exactly six weeks after the first visit. The volunteers' general practitioner and medical specialist (internist or cardiologist) will be informed about their participation. Subjects have to fast for 10 hours before every visit and venous blood samples will be drawn on both visits (a total of 36ml of blood). Subjects will discontinue their usual statin therapy for a period of six weeks. No major risks are involved with temporary discontinuation of statin therapy in stable chronic cardiovascular disease. Volunteers will receive 25 euro's in total for participation. Participation serves to further investigate the relation of statins and potentially beneficial binding of apoB on erythrocytes.

DETAILED DESCRIPTION:
INTRODUCTION:

Previously it has been shown that atherogenic apolipoprotein (apo) B containing lipoproteins bind to erythocytes.1-3 Studies from our laboratory have shown that the binding of apoB on erythrocytes (ery-apoB) may reflect a situation of protection against cardiovascular disease (CVD).4 Mean ery-apoB is significantly lower in subjects with known CVD compared to healthy controls. However, the use of statins could be an important confounding factor, because of its known LDL-C and serum apoB lowering effects.5, 6 In our on-going study population 91% of the patients with CVD were on statin therapy compared to only 19% of the subjects without CVD. Preliminary data showed at least some effect of statin therapy on ery-apoB. A modest, but significant negative correlation was found between ery-apoB and serum apoB and LDL-cholesterol in subjects without statins (Pearson's r -0.172 and -0.185, P < 0.05) but these correlations were lost in subjects using statins. Statins are known for their inhibition of HMG-CoA reductase, which is necessary for the liver to synthesize cholesterol, and increase the expression of hepatic LDL-receptors resulting in lowering of LDL-cholesterol and its related apoB.7, 8 In theory ery-apoB may be lowered by statins as well, which could be an explanation for the differences in ery-apoB between subjects with or without CVD. This interventional study is to explore the effects of statin therapy on ery-apoB.

AIM:

To investigate the effects of statin therapy on plasma levels of erythrocyte-bound apolipoprotein B.

HYPOTHESIS:

Ery-apoB will increase after statin withdrawal due to higher total plasma apoB.

METHODS AND MATERIALS:

Study population Subjects will be males and females aged 18 years or older who are on statin therapy for medical purposes like primary or secondary hypercholesterolemia or the presence of CVD. Exclusion criteria are unstable angina pectoris, an acute cardiovascular event (i.e. myocardial infarction, percutaneous coronary intervention, stroke or bypass surgery) in the last 6 months or the use of any other lipid lowering drug like ezetimibe or fibrates besides statin therapy in the last 6 months.

Study design

A total of 53 subjects will visit the outpatient clinic twice. The following procedures will be performed during the first visit:

* Questionnaire to obtain information about patient's medical history, medication profile and the general practitioners contact information.
* Measurement of anthropometric variables (blood pressure, length, weight and waist).
* Venipuncture (1 Clot tube, 1 Heparin tube, 1 EDTA tube and 1 Glucose tube, a total of 18ml of blood).
* Temporary discontinuation of statin therapy for 6 weeks. Six weeks after the first visit participating subjects will attend the outpatient clinic again for another venipuncture (1 Clot tube, 1 Heparin tube, 1 EDTA tube and 1 Glucose tube, a total of 18ml of blood). Subjects will start again with their original statin therapy afterwards (same type of drug and dosage). However, statin therapy will be initiated earlier if the subject suffers from an acute cardiovascular event during the study period. Study subjects will be monitored by phone for adverse events 8 weeks after finishing the study.

Intervention Statin therapy will be discontinued for a period of six weeks.

Analytical determinations Basic parameters for renal function as well as glucose, CRP, total cholesterol, HDL-C and TG will be determined using Synchrom LX analyzer (Beckman Coulter, Anaheim CA, USA). LDL-C values will be calculated using the Friedewald formula. ApoAI and ApoB will be determined by rate nephelometry using IMAGE by commercially available kits provided by Beckman (Beckman Coulter Anaheim CA, USA). Blood cell counts will be determined automatically using LH analyzer (Beckman Coulter, CA, USA). The leukocyte differentiation will be determined as a five-part differentiation on the same instruments. ApoB on blood cells will be detected by indirect immunofluorescence evaluated by flow cytometry, previously validated and published.9

Required materials

* Flow cytometer (Beckman Coulter, USA)
* Validated measurement protocol for ery-apoB on flow cytometry
* Venous blood drawing equipment and blood tubes
* Funding: Stichting Onderzoek & Ontwikkeling Sint Franciscus Gasthuis and Klinisch Chemisch Laboratorium Sint Franciscus Gasthuis cover the costs

Investigational product The medication group of statins is the product of investigation. The most frequently prescribed statins are simvastatin, atorvastatin, rosuvastatin, pravastatin and fluvastatin with dosages ranging from 5mg to 80mg administered once daily.10 Statins inhibit HMG-CoA reductase, which is necessary for the liver to synthesize cholesterol, and subsequently lowers LDL-cholesterol and its related apo B.7, 8 Atorvastatin and rosuvastatin show the longest terminal half-life (11-14 hours) compared to the other statins (1-3 hours).11 Bioavailability of statins is low due to an extensive first-pass effect intestinally and at the liver and all but pravastatin show active metabolites.11 All active metabolites of statins will be eliminated after discontinuation of statins for six weeks.

Statistics Subjects will serve as their own control group. Therefore, the paired T test will be used to test for significant differences in ery-apoB before and after withdrawal of statin therapy. The differences in ery-apoB before and after withdrawal of statin therapy are checked for normality using the Shapiro-Wilk test. A P-value below 0.05 will be regarded as statistical significant.

Ongoing observational studies have shown a mean difference 0.25 between subjects with and without statin therapy. A recently completed pilot has shown a SD of the difference of 0.64 instead of previously estimated SD of 0.50. To demonstrate a significant difference of ery-apoB with a mean difference of 0.25 a.u. and a SD of the difference of 0.64, at least 53 subjects should be included in the analysis (power is 80%, alpha is 0.05 two-sided).

Safety reporting The investigator will inform the subjects and the reviewing accredited METC if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The study will be suspended pending further review by the accredited METC, except insofar as suspicion jeopardize the subjects' health. The investigator will take care that all subjects are kept informed.

Adverse events (AE) are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigated treatment. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded. A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life threatening, requires hospitalization or prolongation or existing in patients' hospitalization, results in persistent disability of incapacity or affects the safety of the subjects in any way. These serious adverse events will be reported through the web portal "Toetsing Online" to the accredited METC that approved the protocol.

Adverse events that may be expected regarding the withdrawal of statins for a period of six weeks are the occurrence of an acute cardiovascular event or "statin withdrawal syndrome". Studies have shown that discontinuation of statin therapy is associated with worse outcomes after an acute coronary syndrome, stroke or vascular surgery.12 However, no increase in adverse outcomes was observed in patients with stable chronic coronary artery disease following the temporary discontinuation of statin therapy.12 The prevalence of statin related muscle complaints is 1-10%.13 However, the risk of statin related muscle complaints after restarting the statin after withdrawal of four weeks will be very small since study subjects were already on the same statin before participation of the study. There is no clear evidence of any significant harm or effects on quality of life caused by statins in a group of 34.272 study subjects.14

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* use of a statin

Exclusion Criteria:

* use of other lipid lowering drugs, other than statins
* a cardiovascular event in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Apolipoprotein B bound to erythrocytes | 6 weeks
  Change in apollipoprotein B bound to erythrocytes six weeks after cessation of statin therapy

SECONDARY OUTCOMES:
Apolipoprotein B bound to leukocytes | Six weeks
  Change in apolipoprotein B bound to leukocytes after cessation of statin therapy
Leukocyte activation | six weeks
  Change in leukocyte activation markers after cessation of statin therapy:
  * cytoplasmatic MPO in neutrophils
  * CD11b expression on monocytes and neutrophils
  * CD66b expression on neutrophils

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Castro Cabezas, MD, PhD, Study Director — Sint Franciscus Gasthuis
Locations (1):
- Sint Franciscus Gasthuis, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Bovenberg SA, Alipour A, Elte JW, Rietveld AP, Janssen JW, van de Geijn GJ, Njo TN, van Mechelen R, Hervas SM, Cabezas MC. Cell-mediated lipoprotein transport: a novel anti-atherogenic concept. Atheroscler Suppl. 2010 Jun;11(1):25-9. doi: 10.1016/j.atherosclerosissup.2010.04.003. Epub 2010 Apr 27. PMID 20427243
- [Background] Hui DY, Harmony JA. Interaction of plasma lipoproteins with erythrocytes. I. Alteration of erythrocyte morphology. Biochim Biophys Acta. 1979 Feb 2;550(3):407-24. doi: 10.1016/0005-2736(79)90145-7. PMID 217429
- [Background] Hui DY, Noel JG, Harmony JA. Binding of plasma low density lipoproteins to erythrocytes. Biochim Biophys Acta. 1981 Jun 23;664(3):513-26. doi: 10.1016/0005-2760(81)90129-6. PMID 6791697
- [Background] Bovenberg SA, Klop B, Alipour A, Martinez-Hervas S, Westzaan A, van de Geijn GJ, Janssen HW, Njo T, Birnie E, van Mechelen R, Rietveld AP, Elte JW, Castro Cabezas M. Erythrocyte-associated apolipoprotein B and its relationship with clinical and subclinical atherosclerosis. Eur J Clin Invest. 2012 Apr;42(4):365-70. doi: 10.1111/j.1365-2362.2011.02591.x. Epub 2011 Sep 13. PMID 21913916
- [Background] Molgaard J, von Schenck H, Olsson AG. Effects of simvastatin on plasma lipid, lipoprotein and apolipoprotein concentrations in hypercholesterolaemia. Eur Heart J. 1988 May;9(5):541-51. doi: 10.1093/oxfordjournals.eurheartj.a062541. PMID 3402470
- [Background] Bard JM, Luc G, Douste-Blazy P, Drouin P, Ziegler O, Jacotot B, Dachet C, De Gennes JL, Fruchart JC. Effect of simvastatin on plasma lipids, apolipoproteins and lipoprotein particles in patients with primary hypercholesterolaemia. Eur J Clin Pharmacol. 1989;37(6):545-50. doi: 10.1007/BF00562541. PMID 2693115
- [Background] Klop B, Elte JW, Cabezas MC. [Cholesterol homeostasis and enterohepatic connection: new insights in cholesterol absorption]. Ned Tijdschr Geneeskd. 2011;155:A2503. Dutch. PMID 21262010
- [Background] Poli A. Atorvastatin: pharmacological characteristics and lipid-lowering effects. Drugs. 2007;67 Suppl 1:3-15. doi: 10.2165/00003495-200767001-00002. PMID 17910517
- [Background] Alipour A, van Oostrom AJ, Izraeljan A, Verseyden C, Collins JM, Frayn KN, Plokker TW, Elte JW, Castro Cabezas M. Leukocyte activation by triglyceride-rich lipoproteins. Arterioscler Thromb Vasc Biol. 2008 Apr;28(4):792-7. doi: 10.1161/ATVBAHA.107.159749. Epub 2008 Jan 24. PMID 18218988
- [Background] Jukema JW. [The availability of only one statin is inadequate]. Ned Tijdschr Geneeskd. 2005 Dec 10;149(50):2773-4. Dutch. PMID 16385828
- [Background] Garcia MJ, Reinoso RF, Sanchez Navarro A, Prous JR. Clinical pharmacokinetics of statins. Methods Find Exp Clin Pharmacol. 2003 Jul-Aug;25(6):457-81. PMID 12949632
- [Background] Pineda A, Cubeddu LX. Statin rebound or withdrawal syndrome: does it exist? Curr Atheroscler Rep. 2011 Feb;13(1):23-30. doi: 10.1007/s11883-010-0148-x. PMID 21104165
- [Background] Janssen SP, Smulders YM, Gerdes VE, Visseren FL. [Muscle problems due to statins: underestimated]. Ned Tijdschr Geneeskd. 2010;154:A1684. Dutch. PMID 21435278
- [Background] Taylor F, Ward K, Moore TH, Burke M, Davey Smith G, Casas JP, Ebrahim S. Statins for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD004816. doi: 10.1002/14651858.CD004816.pub4. PMID 21249663
- [Derived] de Vries MA, Alipour A, Klop B, van de Geijn GJ, Janssen HW, Njo TL, van der Meulen N, Rietveld AP, Liem AH, Westerman EM, de Herder WW, Cabezas MC. Glucose-dependent leukocyte activation in patients with type 2 diabetes mellitus, familial combined hyperlipidemia and healthy controls. Metabolism. 2015 Feb;64(2):213-7. doi: 10.1016/j.metabol.2014.10.011. Epub 2014 Oct 16. PMID 25456098